CLINICAL TRIAL: NCT05179213
Title: Azacytidine Combined With Chidamide in the Treatment of Relapsed and Refractory Angioimmunoblastic T-cell Lymphoma: a Multicenter Single Arm Phase II Study
Brief Title: Azacytidine Plus Chidamide in the Treatment of Relapsed and Refractory Angioimmunoblastic T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Longfu Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-012
Record Dates: First submitted 2021-12-08; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Angioimmunoblastic T-cell Lymphoma
Keywords: Angioimmunoblastic T-cell Lymphoma; Azacytidine; Chidamide
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — Azacitidine; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Azacytidine combined with chidamide (Experimental): Patients in the experimental arm will received azacytidine plus chidamide treatment. This regimen was repeated every 28 days.
  Interventions: Drug: Azacitidine; Drug: Chidamide

INTERVENTIONS:
Drug: Azacitidine — 75 mg/m2 subcutaneously on days 1-7
Drug: Chidamide — 20mg orally per week continuously

SUMMARY:
This is a multicenter prospective single arm phase II study. The purpose of this study is to evaluate the safety and efficiency of azacytidine combined with chidamide in the treatment of relapsed/refractory angioimmunoblastic T-cell lymphoma.

DETAILED DESCRIPTION:
Azacytidine was given subcutaneously at a dose of 75 mg/m2 on days 1-7. Chidamide was an oral tablet which was administered 20mg twice weekly. This regimen was repeated every 28 days. Treatment was given until disease progression, unacceptable toxicity, or patient/investigator discretion.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed angioimmunoblastic T-cell lymphoma according World Health Organization (WHO) classification;
* Age≥18years;
* ECOG≤2;
* Patients received at least one systemic treatment previously and achieved no remission or relapsed after first-line treatment;
* Adequate bone marrow hematopoietic function: ANC>1.5 × 109/L，HGB>90g/L，PLT>80 × 109/L;
* Adequate organ function: ALT≤3 times ULN, TBil≤1.5 times ULN, SCr≥50ml/min/m2, cardiac function grade 0-2 (NYHA);

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment;
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy;
* Pregnant or lactating women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 1year
  ORR was defined as the proportion of patients who achieved CR or PR as their best response

SECONDARY OUTCOMES:
progression-free survival (PFS) | 1 year
  PFS was defined as time from diagnosis to the date of disease progression or death from any cause or the last follow-up.
Duration of response (DOR) | through study completion, an average of 1 year
  DOR was defined as the time from the first occurrence of CR or PR to the first diagnosis of PD or relapse.
overall survival (OS) | through study completion, an average of 2 year
  OS was defined as time from diagnosis to death from any cause or the last follow-up.
Adverse Events | During the whole treatment
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Dr, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No